CLINICAL TRIAL: NCT07030673
Title: Early Discontinuation of Antibiotic Therapy in Elderly Patients Hospitalized for a Viral Infection
Acronym: ABUSIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); Centre Hospitalier de Beauvais (Other); University Hospital, Caen (Other); Hôpital Les Bateliers, CHU de Lille (Unknown); Centre Hospitalier Roubaix (Unknown); CH SOISSONS (Unknown); Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2023_843_0153
Record Dates: First submitted 2025-03-27; First posted 2025-06-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Elderly; Antibiotics Overuse; Viral Infections; PCR Multiplex
Keywords: viral infections; elderly; antibiotics overuse; PCR multiplex
MeSH Terms: conditions — Virus Diseases | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stop antibiotic (Experimental)
  Interventions: Drug: antibiotic withdrawal
- standard of care (Active Comparator)
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: antibiotic withdrawal — stop antibiotics on viral or negative results
  Arms: stop antibiotic
Drug: Antibiotics — standard of care
  Antibiotics are :
  Amoxicilline-acide clavulanique : 1g x3/j, 7j or Ceftriaxone : 1g/j, 7j or Pipéracilline-Tazobactam : 4g x3/j, 7j or Pristinamycine : 1g x 3/j, 7j
  Arms: standard of care

SUMMARY:
Among winter respiratory viruses, influenza is the most common and therefore responsible for the highest mortality, but parainfluenza and RSV viruses have an even higher risk of mortality (1.6 to 1.9 times), this toll being paid mainly by the elderly and co-morbid population. Futhermore, SARS-Cov2 will probably become endemic and/or epidemic with the same targets of fragile patients. These viral infections are serious, however a bacterial co-infection worsens the prognosis even more: excess risk of mortality = 2.6, 95% CI [1.9-3.7].

Although rare, these co-infections are the subject of a prescription of antibiotics in more than 50% of influenza infections or other serious viral infections. Mainly due to this excess risk of mortality associated with the difficulty of diagnosing these co-infections.

Proper antibiotic use requires preventing this misuse and its harmful consequences in the short and long term at all costs. It is therefore imperative to have solid (grade A) evidence showing that antibiotic therapy in viral infections is not only futile but also potentially harmful.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years affiliated to a social security scheme
* Hospitalized for a lower respiratory infection defined as:

  * the presence of 2 of the following 4 signs:
  * hyperthermia >38°C,
  * hyperleukocytosis ≥12000 or ≤4000,
  * purulent aspirations/sputum,
  * rales on pulmonary auscultation indicating parenchymal damage
  * associated with a pulmonary image (standard X-ray, CT scan or ultrasound)
* Microbiological diagnostic sample taken within 48 hours
* Informed consent of the patient or their representative

Exclusion Criteria:

* Hospitalization planned for < 48 hours or transfer planned to another center within 7 days

  * Patient in septic shock,
  * Febrile aplasia
  * Absence of diagnostic microbiological sampling (> 48 hours after admission)
  * Moribund patient,
  * Death expected within the week
  * Inhalation proven by endoscopy or eyewitness
  * Purulent pleurisy, lung abscess, or other concomitant bacterial infection requiring antibiotic therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of days without antibiotics | day 30

SECONDARY OUTCOMES:
number of side effects of antibiotics | day 30
Mortality at M1 | day 30
martality at day 180 | day 180
Length of hospitalization in acute care | day 30
  Length of hospitalization in acute care (days)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No